CLINICAL TRIAL: NCT03618862
Title: Study of the Effects of Farnesoid X Receptor (FXR) Ligands on the Reactivation of Latent Provirus in Circulating CD4 + T Cells Isolated From Patients With Undetectable HIV Viremia Under cART
Brief Title: Study of the Effects of Farnesoid X Receptor (FXR) Ligands on the Reactivation of Latent Provirus
Acronym: FXReservoir
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0370
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood sampling — Peripheral venous blood collection of 56 mL during a sampling required by routine monitoring of human immunodeficiency virus infection.

SUMMARY:
The Farnesoid X receptor (FXR) is a nuclear receptor that controls the transcription of many genes involved in lipid and glucose metabolism. A recent study opens the hypothesis that Farnesoid X receptor also participates in deoxyribonucleic acid repair mechanisms and possibly in the fight against cell invasion by foreign genomes. This hypothesis implied that modulation of Farnesoid X receptor by ligands could modify Human Immunodeficiency Virus replication. The results of in vitro studies with Human Immunodeficiency Virus-infected cell lines indicate that indeed the modulation of Farnesoid X receptor activity by its ligands induces stimulation of virus production rapidly followed by cell death; the overall effect is therefore antiviral. Farnesoid X receptor ligands have also shown an effect on the reactivation of proviruses in cellular models of viral latency studies. This last data raises the hope of being able to intervene on the reservoir of Human Immunodeficiency Virus.

It is therefore crucial to confirm on quiescent CD4 + T lymphocytes of patients whose viral load is controlled by antiretroviral treatment combining several antiretrovirals the results obtained with the in vitro models.

Providing proof of concept that Farnesoid X receptor agonists can reactivate latent proviruses will open new therapeutic perspectives for attacking the Human Immunodeficiency Virus reservoir with a view to achieving a functional cure for Acquired Immune Deficiency Syndrome. The objective of the study is to confirm ex vivo the data obtained in vitro with cellular models and laboratory viral strains. It is therefore necessary to show that Farnesoid X receptor agonists can reactivate latent viruses or proviruses present in quiescent CD4 + T circulating lymphocytes prepared from venous blood of HIV-positive patients under cART. Human Immunodeficiency Virus-positive patients will be any patients, irrespective of the viral genotype, who initiated antiretroviral therapy, regardless of the combination of antiretrovirals, away from primary infection, when they already had a complete western blot, indicating an evolution of the infection without treatment and constitution of an already evolved reservoir. Patients will have had an undetectable viral load since initiation of treatment with a follow-up of at least one year and will have at least 500 CD4 + T lymphocytes / mm3.

ELIGIBILITY:
Inclusion Criteria:

* human immunodeficiency virus infected patients
* T CD4 > 500/mm3. Viral load undetectable for more than a year under stable treatment. No history of virological failure.
* under first line cART treatment
* Indetectable viral load

Exclusion Criteria:

* Acute or chronic anemias.-
* Acute infections, fever
* Vaccination in the two months preceding inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: human immunodeficiency positive patients under cART.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Reactivation of latent proviruses | 1 day
  The primary endpoint of the study is the presence or absence of reactivation of latent proviruses present in quiescent CD4 + T cells purified from peripheral venous blood following treatment of these cells with Farnesoid X receptor agonists.
  This is a composite endpoint because the reactivation will be determined qualitatively, virus production or not after treatment, and quantitatively, level of production of infectious and / or defective viruses.

CONTACTS AND LOCATIONS:
Locations (1):
- Service des maladies infectieuses et tropicales - Hôpital de la Croix Rousse - GHN, Lyon, France

IPD SHARING:
Plan to Share IPD: No